CLINICAL TRIAL: NCT04524026
Title: RIOTC: Reducing the Impact of Ovarian Stimulation. Novel Approaches to Luteal Support in IVF - Study 2
Brief Title: RIOTC: Reducing the Impact of Ovarian Stimulation. Novel Approaches to Luteal Support in IVF-Study 2
Acronym: RIOTC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nicholas Macklon (Other)
Collaborators: Gedeon Richter Ltd. (Industry); Igenomix (Industry)
Responsible Party: Sponsor-Investigator, Nicholas Macklon, Professor, Zealand University Hospital
Organization: Zealand University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REG-210-2017; 2017-004433-93 (EudraCT Number)
Record Dates: First submitted 2018-09-07; First posted 2020-08-24 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: IVF
Keywords: Letrozole, aromatase inhibitor, luteal phase, IVF
MeSH Terms: interventions — Letrozole; Aromatase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): recFSH and co-treatment with letrozole 5 mg/day from stimulation day 1 on cycle day 2 or 3 until the day before gonadotrophin releasing hormone(GnRH) agonist administration to trigger final oocyte maturation. GnRH antagonist 0.25 mg/day from stimulation day 5 until day of GnRH agonist administration. No luteal phase support.
  Interventions: Drug: Letrozole 5 mg
- Control group (No Intervention): recFSH from stimulation day 1 on cycle day 2 or 3 until the day before GnRH agonist administration to trigger final oocyte maturation. GnRH antagonist 0.25 mg/day from stimulation day 5 until day of GnRH agonist administration. No luteal phase support.

INTERVENTIONS:
Drug: Letrozole 5 mg — recFSH and co-treatment with letrozole 5 mg/day from stimulation day 1 on cycle day 2 or 3 until the day before GnRH agonist administration to trigger final oocyte maturation. GnRH antagonist 0.25 mg/day from stimulation day 5 until day of GnRH agonist administration. No luteal phase support.
  Other Names: Aromatase inhibitor
  Arms: Intervention

SUMMARY:
The goal of the randomised controlled study (RCT) is to identify novel strategies that can improve the luteal phase endocrinology after ovarian stimulation, with the aim of using less or no luteal support in IVF while making the endometrium thinner and more receptive to embryo implantation.

DETAILED DESCRIPTION:
The high estradiol levels generated in IVF by multiple dominant follicles at the follicular-luteal phase transition generate powerful negative feedback at the pituitary gland, effectively switching off gonadotropin production. Without stimulation by endogenous luteinizing hormone (LH), the corpora lutea undergo involution and menstruation follows, preventing the establishment of pregnancy.

To address these detrimental effects of ovarian stimulation, the investigators will do a RCT with the use of aromatase inhibitors, which suppress the conversion of androgens to estrogens to ameliorate the unwanted effects of high estrogens.

This study is designed to test the hypothesis that preventing supra-physiological estrogen levels during ovarian stimulation restricts pituitary suppression sufficiently to allow LH levels to rise and support the corpora lutea, leading to a normal post-ovulatory luteal phase, evidenced by a normal duration and luteal phase endocrine profile. To test this, consenting oocyte donors will be randomized to receive co-treatment with aromatase inhibitors or no co-treatment during ovarian stimulation. Following oocyte retrieval, no luteal support will be provided to donors in both Groups.

ELIGIBILITY:
Inclusion Criteria:

* Meet the clinical criteria for acceptance as oocyte donors (healthy women who volunteers to donate oocytes to other women).
* Regular ovulatory cycle of 26-32 days.
* Age: 18-35 years old.
* Written consent.

Exclusion Criteria:

* Contraindications for ovarian stimulation or aspiration of oocytes according to local guidelines
* Polycystic Ovary Syndrome (PCOS)
* Allergy towards study drug
* Women who have had a hormone or copper intra-uterine device (IUD) within 3 months

Exclusion of patients after earlier inclusion in the study in case of

* Patient withdrawal of consent
* Lack of compliance with medication
* Medical complication arising from IVF treatment that requires the cycle to be terminated
* Serious adverse events (SAE) or serious adverse reactions (SAR) including severe allergy to study drug.
* Specific ARs to study drug: severe degree of hot flushed, severe degree of nausea/vomiting, severe diarrhea, severe degree of muscle and joint pain.

In case of exclusion of a patient after earlier inclusion in the study, a new patient will be included.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Yes, but patients will have genitals examined.
Enrollment: 25 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Length of luteal phase (days from aspiration untill bleeding) | Up to three weeks
  Difference in lengths of days until bleeding (from aspiration until first day of bleeding) of the luteal phase between intervention group and control group.

SECONDARY OUTCOMES:
Phase of endometrial receptivity according to Endometrial Receptivity Array (ERA) test | ERA-test is taken 5 days after aspiration of oocytes.
  Difference in established endometrial tissue and secretion markers of endometrial receptivity between intervention group and controls (genomic profile assessed by ERA test).
Estradiol (E2),progesterone (P), luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels. | Blood samples are taken on 1 day of oocyte aspiration, 2 days after, 5 days after and 14 days after.
  Differences in the area under the curve for plasma E2, P, LH and FSH levels from day of OPU until day 14 post OPU between intervention group and control group.
Endometrium thickness. | Endometrium thickness is measured on 1 day of oocyte aspiration, 2 days after and 5 days after.
  Difference in endometrium thickness 5 days post oocyte pick-up (OPU) between intervention group and controls.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Stephen Macklon, Professor, Principal Investigator — Professor; Marianne Dreyer Holt, MD, Study Director — PhD student
Locations (2):
- Denmark (2):
  - Herlev Hospitals Fertilitetsklinik, Herlev
  - Sjællands Fertilitetsklinik, Køge

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dreyer Holt M, Skouby SO, Bulow NS, Englund ALM, Birch Petersen K, Macklon NS. The Impact of Suppressing Estradiol During Ovarian Stimulation on the Unsupported Luteal Phase: A Randomized Controlled Trial. J Clin Endocrinol Metab. 2022 Aug 18;107(9):e3633-e3643. doi: 10.1210/clinem/dgac409. PMID 35779242